CLINICAL TRIAL: NCT01909297
Title: Comparison of the I-gel, Supreme and Proseal LMA in Paralyzed Patients Undergoing Gynaecological Laparoscopic Surgery With Oropharyngeal Leak Pressure
Brief Title: Comparison of the I-gel, Supreme and Proseal LMA in Paralyzed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mukadder Sanli, assistant professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011/188
Record Dates: First submitted 2013-06-21; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Airway Complication of Anaesthesia
Keywords: airway management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ProSeal LMA (Active Comparator): Supraglottic airway device
  Interventions: Device: PROSEAL LMA
- suprema LMA (Active Comparator): Supraglottic airway device
  Interventions: Device: SUPREMA LMA
- I-gel LMA (Active Comparator): Supraglottic airway device
  Interventions: Device: I-GEL LMA

INTERVENTIONS:
Device: PROSEAL LMA — Size 3,4 or 5 supraglottic device with orogastric drainage tube
  Arms: ProSeal LMA
Device: SUPREMA LMA — Size 3,4 or 5, disposable supraglottic device with orogastric drainage tube
  Arms: suprema LMA
Device: I-GEL LMA — Size 3,4,5 disposable supraglottic device with noninflatable cuff
  Arms: I-gel LMA

SUMMARY:
The investigators aimed to compare of the i-gel, supreme and proseal laryngeal mask airways in paralysed patients undergoing gynaecological laparoscopic surgery with oropharyngeal leak pressure. The investigators also studied their relative ease of insertion, time to insertion and complications of use as secondary outcome measures.

DETAILED DESCRIPTION:
A total of 105 patients scheduled for elective gynaecological laparoscopic procedures in our Inonu University Medical Faculty Hospital were recruited.They were equally randomized into three groups: PLMA, supreme and i-gel groups. All three devices were compared with regard to oropharyngeal leak pressure, number and duration of insertion attempts and complications of airway. Oropharyngeal leak pressure will evaluate including to start,trendelenburg and postoperative at period. Fiberoptic evaluation of the LMA's position were performed after successful insertion and determination of the airway pressures. After one hour patients were evaluated by a blinded independent observer for postoperative complications ( sore throat, dysphonia and dysphagia).

ELIGIBILITY:
Inclusion Criteria:

* 18- 60 YEARS

Exclusion Criteria:

* ASA 3-4 patients
* BMI 40

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change of oropharyngeal leak pressure | 10min, 30 min ,45 min
  During intraoperative period, oropharyngeal leak pressure was measured at three times (10min, 30 min, and 45 min after insertion of devices)

SECONDARY OUTCOMES:
easiness of insertion of the device | 2 min
  During insertion, easiness of the devices were evaluated by a scale

OTHER OUTCOMES:
postoperative complication | 2 hour after operation
  At the second hour of postoperative period, patients will visit and will examine about the complications (sore throat, dysphagia, dysphonia)

CONTACTS AND LOCATIONS:
Overall Officials: mukadder sanli, MD, Principal Investigator — Assistant Prof Dr
Locations (1):
- Inonu University, Malatya, Turkey, Turkey (Türkiye)

REFERENCES:
- [Result] Singh I, Gupta M, Tandon M. Comparison of Clinical Performance of I-Gel with LMA-Proseal in Elective Surgeries. Indian J Anaesth. 2009 Jun;53(3):302-5. PMID 20640137